CLINICAL TRIAL: NCT04959799
Title: Retrospective Observational Study on Dalbavancin Real-life Utilization in Diabetic Patients Suffering From Infections - DALBADIA Study
Brief Title: Dalbavancin Real-life Utilization in Diabetic Patients Suffering From Infections (DALBADIA)
Acronym: DALBADIA
Status: Completed | Type: Observational
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 146(Z)PO20094
Record Dates: First submitted 2021-06-21; First posted 2021-07-13 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Diabetes; Infection
Keywords: Diabetes; ABSSSI; Infection; Gram-positive bacteria; Dalbavancin
MeSH Terms: conditions — Diabetes Mellitus; Infections | interventions — dalbavancin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Dalbavancin — Adult diabetic patients suffering from infections who received the last dose of dalbavancin according to the current standard clinical practice at least 30 (+7) days before enrolment in the study.
  Other Names: Xydalba

SUMMARY:
The study aims to describe the current use of dalbavancin among diabetic patients with infections in a real-world clinical setting in Italy and Spain.

DETAILED DESCRIPTION:
The study aims to describe the current use of dalbavancin in diabetic patients suffering from infections proven or suspected to be caused by Gram-positive or mixed Gram-positive and Gram-negative bacteria (with dalbavancin chosen for treating the Gram-positive component) in Italy and Spain.

As overall strategies to reduce the risk of developing severe infections and poor treatment outcomes among diabetic patients are under-researched and should be explored. This study could increase the knowledge of infection management among diabetic patients treated with dalbavancin in order to support appropriate clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of dalbavancin treatment initiation
* Male and female patients
* Patients who received dalbavancin as targeted or empirical therapy to treat Gram-positive bacterial infection or as anti-Gram-positive component of a treatment regimen for mixed infection (e.g., with concurrent antibacterial or antifungals drugs for covering Gram-negative strains or fungi)
* Patients who received the last dose of dalbavancin according to the current standard clinical practice at least 30 (+7) days before enrolment in the study
* Patients with known type 1 diabetes mellitus (T1DM) or type 2 diabetes mellitus (T2DM) at the time of infectious disease of interest diagnosis
* Patients with available retrospective data in medical charts, including information about dalbavancin treatment and diabetes history
* Patients who gave informed consent and personal data processing consent to take part into the study following local regulation.

Exclusion Criteria:

* Patients enrolled in a clinical trial in which treatment with dalbavancin was managed through a study protocol
* Patients diagnosed with any hyperglycemic state other than T1DM or T2DM at the time of dalbavancin treatment initiation
* Patients with long-term infection (over than 12 months of duration) at the time of dalbavancin treatment initiation
* Previous participation in this study. Participation is defined as having given informed consent in this study
* Pregnant or breast-feeding patients from start time of dalbavancin treatment initiation till enrolment visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult diabetic patients suffering from infections who received the last dose of dalbavancin according to the current standard clinical practice at least 30 (+7) days before enrolment in the study.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Retrospective description of the dalbavancin treatment in diabetic patients. | 4 weeks
  Evidence of dalbavancin treatment choice (number and dates of infusions)
Retrospective description of the utilization of dalbavancin treatment in diabetic patients. | 4 weeks
  Evidence of dalbavancin treatment choice (starting and subsequent dosage)
Retrospective description of the setting of dalbavancin treatment in diabetic patients. | 4 weeks
  Evidence of dalbavancin treatment choice (setting of infusion)

SECONDARY OUTCOMES:
Demographic data | 4 weeks
  Demographic data description (Age and Gender)
Clinical cure of dalbavancin | Up to 8 weeks
  Number of patients with clinical cure evaluated by physicians at end of dalbavancin treatment (i.e., date of last dalbavancin dose administration). Clinical cure is defined as clinical signs and symptoms resolved.
Microbiological success of dalbavancin | Up to 8 weeks
  Number of patients with microbiological success at end of dalbavancin treatment (i.e., date of last dalbavancin dose administration).
  Microbioligical success is defined as culture-confirmed eradication of the Gram-positive pathogens identified at baseline, documented as a negative bacterial culture from the same site as the initial positive baseline culture
Incidence of Adverse Events | Up to 8 weeks
  Safety profile was assessed through the incidence of Adverse Events occurred in patients treated with dalbavancin.

CONTACTS AND LOCATIONS:
Locations (11):
- Italy (6):
  - Ospedale Cardinal Massaia, Asti
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliera Universitaria Policlinico "Paolo Giaccone", Palermo
  - A.O.U. Pisana Presidio Ospedaliero Cisanello, Pisa
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine
  - ASST dei Sette Laghi, Varese
- Spain (5):
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Clinic, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario y Politécnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Morata Ruiz L, Ruggieri A, Falcone M, Pasquau Liano J, Gentile I, Salavert Lleti M, Moreno Nunez L, Cascio A, Tascini C, Loeches Yague M, De Rosa FG, Ori A, Comandini A, Cattaneo A, Grossi PA; DALBADIA study group. Dalbavancin real-life utilization among diabetic patients suffering from infections in Italy and Spain: The DALBADIA retrospective cohort study. J Glob Antimicrob Resist. 2024 Mar;36:200-209. doi: 10.1016/j.jgar.2023.11.015. Epub 2024 Jan 10. PMID 38211660